CLINICAL TRIAL: NCT00727051
Title: Comparison of Coronary CT Angiography With Conventional Coronary Angiography in Liver and Lung Transplant Candidates.
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H9730-30837
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: invasive coronary angiography; multidetector coronary CTA; coronary artery disease; detecting coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Liver and lung transplant candidates referred for coronary angiography will be invited to participate in the study.

SUMMARY:
The overall goal of this study is to determine if non-invasive imaging with state of the art CT coronary angiography can be used to screen for coronary artery disease in high risk patients prior to liver and lung transplantation. The current protocol for coronary artery disease assessment at UCSF before liver and lung transplantation involves screening with stress tests and/or coronary angiograms in patients with increased risk of coronary artery disease. Coronary angiogram will be used as gold standard for assessment of coronary CTA accuracy.

ELIGIBILITY:
Inclusion Criteria:

1. Liver transplant candidates referred for invasive coronary angiography which include:

   * Patients with suspicious symptoms for CAD or;
   * Asymptomatic patients;
   * Abnormal non-invasive testing or 1 major risk factor for coronary artery disease or LVEF < 60% on echo.
2. Lung transplant candidates referred for invasive coronary angiography which include:

   * Patients with suspicious symptoms for CAD or;
   * Asymptomatic patients;
   * Abnormal non-invasive testing or 1 major risk factor for coronary artery disease or LVEF < 60% on echo in patients with low SVR (typical for ESLD).
3. Any ethnic background is acceptable.

Exclusion Criteria:

1. Patients with contraindications for the use of iodinated contrast (allergic reaction, renal failure, multiple myeloma, etc) will be excluded.
2. Children and pregnant women will be excluded because of risks associated with radiation exposure.
3. Patients must have no atrial fibrillation, as this will interfere with cardiac gating for the examination.
4. Patients unable to give informed consent will be excluded as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver and lung transplant candidates referred for coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
patients suspected of having coronary artery disease (CAD) | 1-30 days before invasive coronary angiography is performed

CONTACTS AND LOCATIONS:
Overall Officials: Karen G Ordovas, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Zoghbi GJ, Patel AD, Ershadi RE, Heo J, Bynon JS, Iskandrian AE. Usefulness of preoperative stress perfusion imaging in predicting prognosis after liver transplantation. Am J Cardiol. 2003 Nov 1;92(9):1066-71. doi: 10.1016/j.amjcard.2003.06.003. PMID 14583357
- [Background] Findlay JY, Keegan MT, Pellikka PP, Rosen CB, Plevak DJ. Preoperative dobutamine stress echocardiography, intraoperative events, and intraoperative myocardial injury in liver transplantation. Transplant Proc. 2005 Jun;37(5):2209-13. doi: 10.1016/j.transproceed.2005.03.023. PMID 15964381
- [Background] Davidson CJ, Gheorghiade M, Flaherty JD, Elliot MD, Reddy SP, Wang NC, Sundaram SA, Flamm SL, Blei AT, Abecassis MI, Bonow RO. Predictive value of stress myocardial perfusion imaging in liver transplant candidates. Am J Cardiol. 2002 Feb 1;89(3):359-60. doi: 10.1016/s0002-9149(01)02244-5. No abstract available. PMID 11809445
- [Background] Snell GI, Richardson M, Griffiths AP, Williams TJ, Esmore DS. Coronary artery disease in potential lung transplant recipients > 50 years old: the role of coronary intervention. Chest. 1999 Oct;116(4):874-9. doi: 10.1378/chest.116.4.874. PMID 10531146
- [Background] Kaza AK, Dietz JF, Kern JA, Jones DR, Robbins MK, Fiser SM, Long SM, Bergin JD, Kron IL, Tribble CG. Coronary risk stratification in patients with end-stage lung disease. J Heart Lung Transplant. 2002 Mar;21(3):334-9. doi: 10.1016/s1053-2498(01)00387-4. PMID 11897521
- [Background] Ben-Dor I, Shitrit D, Kramer MR, Iakobishvili Z, Sahar G, Hasdai D. Is routine coronary angiography and revascularization indicated among patients undergoing evaluation for lung transplantation? Chest. 2005 Oct;128(4):2557-62. doi: 10.1378/chest.128.4.2557. PMID 16236923
- [Background] Herzog C, Britten M, Balzer JO, Mack MG, Zangos S, Ackermann H, Schaechinger V, Schaller S, Flohr T, Vogl TJ. Multidetector-row cardiac CT: diagnostic value of calcium scoring and CT coronary angiography in patients with symptomatic, but atypical, chest pain. Eur Radiol. 2004 Feb;14(2):169-77. doi: 10.1007/s00330-003-2197-9. Epub 2003 Dec 20. PMID 14689229
- [Background] Leschka S, Alkadhi H, Plass A, Desbiolles L, Grunenfelder J, Marincek B, Wildermuth S. Accuracy of MSCT coronary angiography with 64-slice technology: first experience. Eur Heart J. 2005 Aug;26(15):1482-7. doi: 10.1093/eurheartj/ehi261. Epub 2005 Apr 19. PMID 15840624
- [Background] Raff GL, Gallagher MJ, O'Neill WW, Goldstein JA. Diagnostic accuracy of noninvasive coronary angiography using 64-slice spiral computed tomography. J Am Coll Cardiol. 2005 Aug 2;46(3):552-7. doi: 10.1016/j.jacc.2005.05.056. PMID 16053973
- [Background] Pannu HK, Alvarez W Jr, Fishman EK. Beta-blockers for cardiac CT: a primer for the radiologist. AJR Am J Roentgenol. 2006 Jun;186(6 Suppl 2):S341-5. doi: 10.2214/AJR.04.1944. PMID 16714607